CLINICAL TRIAL: NCT04608721
Title: Effects of Postpartum Anxiety on Breastfeeding and Infant Health Among Taiwanese Women: a Longitudinal Study
Brief Title: Postpartum Anxiety, Breastfeeding and Infant Health Among Taiwanese Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology, Taiwan (Other Government)
Collaborators: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Yuh-Kae Shyu, Assistant Professor, Ministry of Science and Technology, Taiwan
Other Study IDs: 109-FJUH-12
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Postpartum Anxiety; Breastfeeding; Infant Conditions
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postpartum Anxiety: Postpartum anxiety will be assessed at 1-3 days (T1), 1(T2), 3 (T3), 6 (T4) and 12 months (T5) postpartum by using the State-Trait Anxiety Inventory (STAI).
  Interventions: Other: Postpartum Anxiety

INTERVENTIONS:
Other: Postpartum Anxiety — Postpartum anxiety will be assessed at 1-3 days (T1), 1(T2), 3 (T3), 6 (T4) and 12 months (T5) postpartum by using the State-Trait Anxiety Inventory (STAI) with a score ≥40 serving as a positive screen.
  Other Names: PPA

SUMMARY:
This is a prospective, longitudinal and observational study designed to investigate the trajectories of postpartum anxiety and its determinants in the first year after childbirth. This study also examine the associations between postpartum anxiety and infant health outcome, including breastfeeding patterns, excessive crying and body weight growth. Primipara aged 20-49 with term baby will be invited. Demographics, maternal-newborn characteristics, and anxiety symptoms will be collected during the first week postpartum (T1). Questionnaires will be follow-up by mail and telephone reminder in 1 (T2), 3 (T3), 6 (T4) and 12 months (T5) postpartum. The primary outcome is postpartum anxiety using the Spielberger's State-Trait Anxiety Inventory (STAI); the secondary outcomes are infant health outcomes including breastfeeding patterns, excessive crying and body weight growth. A linear mixed model (LMM) is used to determine the trajectories of postpartum anxiety over time and to examine whether specific demographic and maternal characteristics predict the trajectories of postpartum anxiety. The key findings may contribute to promote early identification and secondary preventive interventions for women with postpartum anxiety.

DETAILED DESCRIPTION:
Ditto

ELIGIBILITY:
Inclusion Criteria:

* 20-49 years old
* Primipara

Exclusion Criteria:

* Preterm birth
* Infants with severe congenital malformations/medical conditions or Fetal/neonatal death
* Current use of antidepressant or antipsychotics
* Thoughts of self-harm or suicide

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects will be recruited in 1-3 days postpartum from the birth center or the postpartum ward in the hospitals in northern Taiwan. The well-trained research assistant/registered nurse, responsible for data collection, recognized potential subjects from their medical records, contacted the women and after explaining the aim of study, invited them to complete the baseline questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Postpartum anxiety | Baseline
  Assessments using the Spielberger's State-Trait Anxiety Inventory (STAI) for self-reported anxiety symptoms
Postpartum anxiety | One month from baseline
  Assessments using the Spielberger's State-Trait Anxiety Inventory (STAI) for self-reported anxiety symptoms
Postpartum anxiety | Three months from baseline
  Assessments using the Spielberger's State-Trait Anxiety Inventory (STAI) for self-reported anxiety symptoms
Postpartum anxiety | Six months from baseline
  Assessments using the Spielberger's State-Trait Anxiety Inventory (STAI) for self-reported anxiety symptoms
Postpartum anxiety | Twelve months from baseline
  Assessments using the Spielberger's State-Trait Anxiety Inventory (STAI) for self-reported anxiety symptoms

SECONDARY OUTCOMES:
Infant health outcomes | Baseline
  Including breastfeeding patterns, excessive crying and body weight growth
Infant health outcomes | One month from baseline
  Including breastfeeding patterns, excessive crying and body weight growth
Infant health outcomes | Three months from baseline
  Including breastfeeding patterns, excessive crying and body weight growth
Infant health outcomes | Six months from baseline
  Including breastfeeding patterns, excessive crying and body weight growth
Infant health outcomes | Twelve months from baseline
  Including breastfeeding patterns, excessive crying and body weight growth

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Kae Shyu, Principal Investigator — Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University, New Taipei City, Xinzhuang Dist, Taiwan